CLINICAL TRIAL: NCT06779630
Title: A Prospective Multicenter Single Arm Study to Assess the Safety and Effectiveness of the Orsiro Mission 48-mm Sirolimus-Eluting Coronary Stent System for the Treatment of Subjects With Atherosclerotic Lesion(s)
Brief Title: Safety and Effectiveness of the Orsiro Mission 48-mm Sirolimus Eluting Coronary Stent System in Subjects With Coronary Artery Lesions
Acronym: BIOFLOW-48
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teleflex (Industry)
Collaborators: BIOTRONIK AG (A Teleflex Company) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G240288
Record Dates: First submitted 2025-01-14; First posted 2025-01-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: Orsiro Mission; Sirolimus-Eluting; Coronary Stent System; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Orsiro Mission 48-mm Sirolimus-Eluting Coronary Stent System (Experimental)
  Interventions: Device: Orsiro Mission 48-mm Sirolimus-Eluting Coronary Stent System

INTERVENTIONS:
Device: Orsiro Mission 48-mm Sirolimus-Eluting Coronary Stent System — Orsiro Mission is composed of a device (coronary stent system including a cobalt chromium stent platform) and a drug product (a formulation of sirolimus) contained in a bioabsorbable polymer coating.

SUMMARY:
The purpose of the study is to assess the safety and efficacy of the Orsiro® Mission 48- mm Sirolimus-Eluting Coronary Stent System in the treatment of subjects with atherosclerotic lesion(s) >36 mm and ≤ 44 mm in length (by visual estimate) in the native coronary arteries with a reference vessel diameter of 2.25 mm to 4.0 mm.

Patients enrolled in the United States will be followed for 2 years post index procedure with follow-up visits at 1, 6, 12 months and 2 years post index procedure. Patients enrolled outside of the United States will be followed through 5 years post index procedure with additional follow-up visits at 3 and 5 years post index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age
2. Subject is able to understand the nature of the study and provide written informed consent.

   For sites outside of the United States: Note: For subjects presenting with STEMI and not in a position to read, interpret and sign the informed consent form, oral informed consent is required.
3. Subject is an acceptable candidate for percutaneous coronary intervention (PCI) according to the applicable guidelines.
4. Subject is an acceptable candidate for CABG.
5. Subject is eligible for dual antiplatelet therapy (DAPT) according to guidelines.
6. Subject has clinical evidence of ischemic heart disease, stable or unstable angina pectoris or documented silent ischemia.
7. Subject is willing and able to comply with study follow-up requirements.

Angiographic inclusion criteria:

1. Subject has only one target lesion in a native coronary artery to be treated with the investigational device.

   Note: One additional non-target lesion may be treated with a non-investigational treatment (e.g. stent, balloon angioplasty, atherectomy) with the exception of brachytherapy, if it is located in a different coronary artery. The non-target lesion must be treated first and must be deemed an angiographic success. (Angiographic success is defined by a residual diameter stenosis < 30% with TIMI 3 flow, as visually assessed by the physician, without the presence of prolonged chest pain or ECG changes consistent with MI.)

   Note: Multiple focal stenoses will be considered as a single lesion if they are amenable to treatment with a single study device.
2. Target lesion must be > 36 mm and ≤ 44 mm in length by operator visual estimate and must be amenable to treatment with a single study device.
3. Target vessel must have a reference vessel diameter of 2.25-4.0 mm by operator visual estimate.
4. For sites in United States: Target lesion must be de novo or restenotic lesion in native coronary artery; restenotic lesion must have been treated with a standard PTCA only.

   For sites outside of the United States: Target lesion can be de novo, restenotic or in-stent restenotic, and must be located in a native coronary artery.
5. Target lesion must have angiographic evidence of ≥ 50% and < 100% stenosis (by operator visual estimate which may be assisted by QCA / IVUS / OCT). Target lesion stenosis < 70% should have clinical justification for treatment as per local standards.
6. Target vessel must have a Thrombolysis In Myocardial Infarction (TIMI) flow > 1.

For sites outside of the United States: Note: For STEMI, TIMI flow > 1 prior to stent implantation (after opening the vessel with a guide wire or a balloon).

Exclusion Criteria:

1. For sites in United States only: Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute ST elevation myocardial infarction (STEMI) within 72 hours prior to the index procedure.

   Note: Hemodynamically stable non-STEMI (NSTEMI) subjects are eligible for study enrollment.
2. Subject is hemodynamically unstable.
3. Subject is pregnant and/or breastfeeding or intends to become pregnant during the duration of the study.
4. Subject has a known allergy to contrast medium that cannot be adequately pre-medicated, or any known allergy to thienopyridine, aspirin, both heparin and bivalirudin, L-605 cobalt-chromium (Co-Cr) alloy or one of its major elements (cobalt, chromium, tungsten and nickel), acrylic, fluoropolymers, silicon carbide, PLLA or sirolimus.
5. Revascularization of any target vessel within 12 months prior to the index procedure or previous PCI of any non-target vessel within <72 hours prior to the index procedure.
6. Future planned PCI (including staged procedure) or CABG after the index procedure.
7. Planned surgery or dental surgical procedure within 6 months of index procedure unless dual antiplatelet therapy can be maintained throughout the peri-surgical period.
8. History of a stroke or transient ischemic attack (TIA) within 6 months prior to the index procedure.
9. Subjects with active bleeding disorders, active coagulopathy, or any other reason, who are ineligible for DAPT.
10. Subject will refuse blood transfusions.
11. Subject has a left ventricular ejection fraction (LVEF) < 30% within 6 months prior to or during the index procedure that was documented by any method.
12. Subject is dialysis dependent or has impaired renal function (i.e., serum creatinine > 2.5 mg/dL or 221 µmol/L, determined within 7 days prior to the index procedure).
13. Subject has a documented white blood cell count < 3,000 white blood cells/mm3 or a documented platelet count < 100,000 platelets/mm3 or > 700,000 platelets/mm3.
14. Subject is receiving oral or intravenous immunosuppressive therapy (inhaled steroids are permitted) or has known life-limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus; diabetes mellitus is permitted).
15. Subject is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure or has a malignancy that is not in remission.
16. Subjects under oral anticoagulation therapy (OAC) prior to index procedure unless DAPT + OAC (i.e. triple therapy) can be maintained according to guidelines.
17. Subject has life expectancy of < 1 year.
18. Subject is currently participating or plans to participate in another clinical investigation with an investigational device or an investigational drug.
19. In the investigator's opinion, subject will not be able to comply with the follow-up requirements.

Angiographic exclusion criteria:

1. Target lesion is excluded if it meets any of the following criteria:

   1. Lesion is located within or treated through a saphenous vein graft or arterial graft.
   2. Lesion location is within the left main coronary artery.
   3. Lesion location is within 3 mm of the origin of the left anterior descending (LAD) or left circumflex (LCX) coronary arteries.
   4. Involves a side branch of > 2.0 mm in diameter that requires a two-device strategy after pre-dilatation.
   5. Lesion is totally occluded (100% stenosis).
   6. For sites in United States only: Lesion is a restenotic lesion that was previously treated with a bare metal or drug eluting stent (in-stent restenosis).
2. Target vessel/lesion is excessively tortuous/angulated or is severely calcified, that would prevent complete inflation of an angioplasty balloon. This assessment should be based on visual estimation.
3. Site sites in the United States: Target vessel has angiographic evidence of thrombus.

   For sites outside of the United States: Target vessel has angiographic evidence of unresolved large thrombus burden despite of thrombus aspiration.

   Note: Thrombus aspiration is left at the discretion of the implanting physician.
4. Target vessel was treated with brachytherapy any time prior to the index procedure.
5. Unsuccessful target lesion pre-dilatation, defined as residual stenosis > 50% (by visual estimation) and/or angiographic complications (e.g., distal embolization, side branch closure, dissection greater than National Heart, Lung, Blood Institute type C), and/or, for sites outside of the United States, coronary aneurysms.
6. Non-target lesion is excluded if it meets any of the following criteria:

   1. Any of the target lesion angiographic exclusion criteria except for 1c
   2. Lesion is located within the target vessel.
   3. Lesion is > 36 mm by operator visual estimate.
   4. Lesion requires additional, unplanned stents to treat a complication.
   5. Lesion treatment is not deemed an angiographic success. (Angiographic success is defined by a residual diameter stenosis < 30% with TIMI 3 flow, as visually assessed by the physician, without the presence of prolonged chest pain or ECG changes consistent with MI.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) rate at 12 months post-index procedure | 12 months
  The primary endpoint will be target lesion failure (TLF) rate at 12 months post-index procedure. TLF is defined as a composite of cardiac death, target vessel Q-wave or non-Q-wave myocardial infarction (TV-MI), or clinically driven target lesion revascularization (CD-TLR).

SECONDARY OUTCOMES:
Device success | Hospital Discharge (6-24 hours post-index procedure)
  Device success, defined as attainment of < 30% residual stenosis of the target lesion (based on operator visual estimate) using the Orsiro Mission study stent only.
Procedure success | Hospital Discharge (6-24 hours post-index procedure)
  Procedure success, defined as attainment of < 30% residual stenosis of the target lesion (based on operator visual estimate) using the Orsiro Mission study stent only without occurrence of in-hospital major adverse cardiac events (MACE).
All-cause death | 1, 6, 12 months and 2, 3, and 5 years post-index procedure
Any myocardial infarction (MI) | 1, 6, 12 months and 2, 3, and 5 years post-index procedure
Cardiac death or myocardial infarction (MI) | 1, 6, 12 months and 2, 3, and 5 years post-index procedure
Major cardiac adverse events (MACE) and individual MACE components | 1, 6, 12 months and 2, 3, and 5 years post-index procedure
  MACE is defined as a composite of all-cause death, Q-wave or non-Q-wave MI, and any clinically driven target lesion revascularization (TLR).
Target lesion failure (TLF) and individual TLF components | 1, 6, 12 months and 2, 3, and 5 years post-index procedure
  TLF is defined as a composite of cardiac death, target vessel Q-wave or non-Q-wave myocardial infarction (TV-MI), or clinically driven target lesion revascularization (CD-TLR).
Target vessel failure (TVF) and individual TVF components | 1, 6, 12 months and 2, 3, and 5 years post-index procedure
  TVF is defined as a composite of cardiac death, target vessel Q-wave or non-Q-wave myocardial infarction (TV-MI), and clinically driven target vessel revascularization (CD-TVR).
Target lesion revascularization (TLR) | 1, 6, 12 months and 2, 3, and 5 years post-index procedure
Target vessel revascularization (TVR) | 1, 6, 12 months and 2, 3, and 5 years post-index procedure
Stent thrombosis | 1, 6, 12 months and 2, 3, and 5 years post-index procedure
  Stent thrombosis will be assessed according to Academic Research Consortium - 2 (ARC-2) definitions.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (4):
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Baylor Scott & White The Heart Hospital - Dallas, Dallas, Texas
  - Ascension Texas Cardiovascular, Kyle, Texas
  - Charleston Area Medical Center, Charleston, West Virginia
- Austria (2):
  - Klinische Abteilung für Kardiologie, Medizinische Universität Graz, Graz, Styria
  - Universitätsklinik für Innere Medizin II, Klinische Abteilung für Kardiologie, Medizinische Universität Wien, Vienna, Vienna
- Institut Arnault Tzanck, Saint-Laurent-du-Var, Provence-Alpes-Côte d'Azur Region, France
- Germany (3):
  - Universitätsklinikum Mannheim, I. Medizinische Klinik, Mannheim, Baden-Wurttemberg
  - Klinikum Fürth, Fürth, Bavaria
  - Segeberger Kliniken GmbH, Bad Segeberg, Schleswig-Holstein
- Miedziowe Centrum Zdrowia SA, Lubin, Lower Silesian Voivodeship, Poland
- Switzerland (2):
  - University hospital Basel, Basel, Canton of Basel-City
  - Istituto Cardiocentro Ticino, Lugano, Canton Ticino

IPD SHARING:
Plan to Share IPD: No
No IPD sharing is planned at this time. This study evaluates an investigational device under an FDA IDE. The sponsor may consider sharing de-identified IPD under controlled access following completion of primary endpoint analysis and regulatory review. Summary results will be reported in scientific publications and public registries.